CLINICAL TRIAL: NCT00642447
Title: Helium:Oxygen Versus Air:Oxygen Nonivasive Positive Pressure Ventilation in Patients Exposed to Sulfur Mustard
Brief Title: Helium:Oxygen Noninvasive Positive Pressure Ventilation in Patients Exposed to Sulfur Mustard
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: B12406
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Last update posted 2008-03-25 (Estimated); Status verified 2008-03

CONDITIONS: Bronchiolitis; Chronic Bronchitis
Keywords: noninvasive ventilation; helium; oxygen; sulfur mustard; chronic bronchitis; bronchiolitis
MeSH Terms: conditions — Bronchiolitis; Bronchitis, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: helium:oxygen mixture

INTERVENTIONS:
Drug: helium:oxygen mixture

SUMMARY:
to assess the effect of Heliox with Noninvasive positive pressure ventilation to decrease dyspnea and improve physiologic and respiratory measures in patients with a previous exposure to Sulfur Mustard gas.

ELIGIBILITY:
Inclusion Criteria:

* exposure to sulfur mustard
* worsening dyspnea during the last 10 days
* respiratory rate of >25/min
* arterial pH<7.35
* PaCO2 of >50 mmHg
* PaO2 of <50 mmHg

Exclusion Criteria:

* recent pneumothorax (<1 month)
* severe respiratory failure or hemodynamic instability with forthcoming intubation
* FIO2 of <0.4
* impaired consciousness or absence of patient cooperation
* facial lesions precluding NIPPV

Ages: 38 Years to 59 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23
Dates: Start 2007-04

CONTACTS AND LOCATIONS:
Locations (1):
- BMSU, Tehran, Tehran Province, Iran